CLINICAL TRIAL: NCT00489827
Title: Phase III Study of Intravenous Glutamate Infusion for Metabolic Protection of the Heart in Surgery for Unstable Coronary Artery Disease
Brief Title: Glutamate for Metabolic Intervention in Coronary Surgery
Acronym: GLUTAMICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Region Örebro County (Other); Blekingesjukhuset, Karlskrona (Unknown)
Responsible Party: Principal Investigator, Rolf Svedjeholm, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 151:2003/70403; 20030595 (Registry Identifier: 151/2003/70403 Swedish Medical Product Agency)); M76-05 (Other: Regional Ethical Review Board in Linkoping)
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Bypass; Myocardial Ischemia; Myocardial Infarction; Coronary Artery Disease
Keywords: Coronary Artery Bypass; Myocardial Protection; Angina, Unstable; Myocardial Ischemia; Myocardial Infarction; Unstable Coronary Artery Disease; Glutamate
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Coronary Artery Disease; Angina, Unstable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous glutamate (Active Comparator): Intravenous infusion of 0.125 M glutamic acid solution at a rate of 1.65 ml/hour and kg body weight beginning with institution of anesthesia and stopping 2 hours after unclamping of aorta in patients operated for unstable coronary artery disease.
  Interventions: Other: Intravenous glutamate infusion
- Saline infusion (Placebo Comparator): Intravenous infusion of saline at a rate of 1.65 ml/hour and kg body weight beginning with institution of anesthesia and stopping 2 hours after unclamping of aorta in patients operated for unstable coronary artery disease.
  Interventions: Drug: Intravenous infusion of saline

INTERVENTIONS:
Drug: Intravenous infusion of saline — Intravenous infusion of isotonic saline at a rate of 1.65 ml/hour and kg body weight beginning with institution of anesthesia and stopping 2 hours after unclamping of aorta in patients operated for unstable coronary artery disease.
  Arms: Saline infusion
Other: Intravenous glutamate infusion — Intravenous infusion of 0.125 M glutamic acid solution at a rate of 1.65 ml/hour and kg body weight beginning with institution of anesthesia and stopping 2 hours after unclamping of aorta in patients operated for unstable coronary artery disease.
  Arms: Intravenous glutamate

SUMMARY:
The main purpose of this study is to determine whether intravenous glutamate infusion given in association with surgery for unstable coronary artery disease can protect the heart from myocardial injury, postoperative heart failure and death.

DETAILED DESCRIPTION:
Myocardial preservation in cardiac surgery has mainly focused on the period when the heart is arrested (cross-clamp time). Today the heart can be arrested for up to 2-3 hours without major consequences. However, in spite of comparatively short cross-clamp times approximately 10% of the patients undergoing coronary surgery sustain significant myocardial injury whereas perioperative myocardial infarction is rare in aortic valve surgery despite longer cross-clamp times. The reason for this is that preoperative ischemia, and to some extent postoperative ischemia, remain major risk factors for development of myocardial infarction in patients with ischemic heart disease. In light of this, we suggest that efforts to improve outcome and reduce permanent myocardial damage should focus on the preoperative and the postoperative phase of coronary surgery. Furthermore, efforts should be instituted to reduce reperfusion injury and minimize permanent myocardial damage in long-standing or severe myocardial ischemia.

Metabolic intervention with intravenous glutamate infusion, offers the prospect of addressing the issues above and extending myocardial protection into the pre- and postoperative phase. Glutamate is an important substrate for the intermediary metabolism of the heart, particularly in association with ischemia. The effects of glutamate are partly related to its role in the malate-aspartate shuttle, transporting reducing equivalents across the mitochondrial membrane, regulating the NAD/NADH balance in the cytosol of the cells, and thereby enhancing anaerobic glycolysis during ischemia. Furthermore, glutamate contributes to an alternative anaerobic pathway for regeneration of high-energy phosphates, by substrate level phosphorylation in the Krebs cycle. Glutamate also improves clearance of metabolic waste produced during ischemia such as lactate and NH3, by taking part in the reactions involving transamination of pyruvate to alanine and of glutamate to glutamine. During reperfusion glutamate contributes to the replenishment of Krebs cycle intermediates lost during ischemia, which is essential for recovery of oxidative metabolism.

Administration of glutamate to patients with stable angina pectoris has been found to increase tolerance to stress-induced ischemia. Ischemia before onset of cardiopulmonary bypass has been established as a major risk factor for postoperative myocardial infarction. Patients with unstable coronary artery disease may have critical ischemia at rest and are particularly vulnerable to the increased oxygen demands during the early stages of coronary surgery. In a pilot study on patients operated urgently for unstable angina we found metabolic signs compatible with improved tolerance to ischemia before surgery and improved recovery of oxidative metabolism during early reperfusion. These results warrant further studies to evaluate the potential clinical benefit of preoperative glutamate infusion extended into the early postoperative period.

Comparisons: Intravenous infusion of 0.125 M glutamic acid solution v saline at a rate of 1.65 ml/hour and kg body weight beginning with institution of anesthesia and stopping 2 hours after unclamping of aorta in patients operated for unstable coronary artery disease.

Preliminary power analysis (80% power; p<0.05) suggests that 2214 patients will be required with regard to primary end-point assuming 30% reduction of events occurring in 12% of untreated patients.

Stage I of the study comprises 800 patients* and will lead to an interim analysis with report of secondary end-points** and recalculation of sample-size with regard to primary end-point. An adaptive design with regard to primary end-point and analysis performed by external statistician blinded to the investigators will be used to avoid increasing the risk for type I error.

*Patient number 800 is anticipated to be enrolled during the summer of 2009 and for practical reasons all patients enrolled until the end of August 2009 will comprise the interim analysis.

**Secondary end-points include analysis of markers for myocardial injury (CK-MB, troponin-T), markers for hemodynamic adequacy (mixed venous oxygen saturation), renal function (p-creatinine, p-Cystatin C), brain injury (S100B, clinical signs). As a substudy a blinded analysis of the value of NT-pro BNP (obtained immediately before surgery, 24 hours postoperatively and on the 3rd postoperative day) as marker of postoperative heart failure and outcome will be conducted. NT-pro BNP will also be related to treatment with glutamate or placebo. Similar evaluation will involve markers troponin-T, p-Cystatin C and mixed venous oxygen saturation. For further details see outcome measures.

Substudies will involve subgroup analyses of patients with regard to combined CABG + valve procedures, severely unstable patients requiring emergency surgery / intravenous nitrates, preoperative LV-dysfunction and patients with diabetes. For further details see outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* surgery for unstable coronary artery disease (unstable angina, non-STEMI)
* accepted for surgery < 2 weeks after STEMI
* coronary surgery for indications above performed with or without cardiopulmonary bypass
* coronary surgery for indications above with or without simultaneous valve procedure

Exclusion Criteria:

* informed consent not possible because of critical condition or other reason
* preoperative use of inotropes or mechanical circulatory assist
* preoperative dialysis
* redo-procedure
* unexpected intraoperative finding / event that increased the dignity of the procedure to overshadow the originally planned operation
* body weight > 125 kg
* food allergy known to have caused flush, rash or asthma

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2005-10; Primary Completion 2009-12 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Svedjeholm, MD PhD, Study Director — University Hospital, Linkoeping
Locations (3):
- Sweden (3):
  - Blekingesjukhuset, Karlskrona, Karlskrona
  - University Hospital, Linköping, Linköping
  - University Hospital, Örebro, Örebro

REFERENCES:
- [Background] Slogoff S, Keats AS. Does perioperative myocardial ischemia lead to postoperative myocardial infarction? Anesthesiology. 1985 Feb;62(2):107-14. doi: 10.1097/00000542-198502000-00002. PMID 3970360
- [Background] Dahlin LG, Olin C, Svedjeholm R. Perioperative myocardial infarction in cardiac surgery--risk factors and consequences. A case control study. Scand Cardiovasc J. 2000 Oct;34(5):522-7. doi: 10.1080/140174300750064710. PMID 11191945
- [Background] Mudge GH Jr, Mills RM Jr, Taegtmeyer H, Gorlin R, Lesch M. Alterations of myocardial amino acid metabolism in chronic ischemic heart disease. J Clin Invest. 1976 Nov;58(5):1185-92. doi: 10.1172/JCI108571. PMID 993339
- [Background] Thomassen AR, Nielsen TT, Bagger JP, Henningsen P. Myocardial exchanges of glutamate, alanine and citrate in controls and patients with coronary artery disease. Clin Sci (Lond). 1983 Jan;64(1):33-40. doi: 10.1042/cs0640033. PMID 6129934
- [Background] Pisarenko OI, Baranov AV, Aleshin OI, Studneva IM, Pomerantsev EA, Nikolaeva LF, Savchenko AP, Pavlov NA. Features of myocardial metabolism of some amino acids and ammonia in patients with coronary artery disease. Eur Heart J. 1989 Mar;10(3):209-17. doi: 10.1093/oxfordjournals.eurheartj.a059468. PMID 2707269
- [Background] Thomassen A, Botker HE, Nielsen TT, Thygesen K, Henningsen P. Effects of glutamate on exercise tolerance and circulating substrate levels in stable angina pectoris. Am J Cardiol. 1990 Jan 15;65(3):173-8. doi: 10.1016/0002-9149(90)90080-k. PMID 1967510
- [Background] Thomassen A, Nielsen TT, Bagger JP, Pedersen AK, Henningsen P. Antiischemic and metabolic effects of glutamate during pacing in patients with stable angina pectoris secondary to either coronary artery disease or syndrome X. Am J Cardiol. 1991 Aug 1;68(4):291-5. doi: 10.1016/0002-9149(91)90821-2. PMID 1858669
- [Background] Thomassen AR. Myocardial uptake and effects of glutamate during non-ischaemic and ischaemic conditions. A clinical study with special reference to possible interrelationships between glutamate and myocardial utilization of carbohydrate substrates. Dan Med Bull. 1992 Dec;39(6):471-88. No abstract available. PMID 1361429
- [Background] Beyersdorf F, Kirsh M, Buckberg GD, Allen BS. Warm glutamate/aspartate-enriched blood cardioplegic solution for perioperative sudden death. J Thorac Cardiovasc Surg. 1992 Oct;104(4):1141-7. PMID 1405674
- [Background] Pisarenko OI, Portnoy VF, Studneva IM, Arapov AD, Korostylev AN. Glutamate-blood cardioplegia improves ATP preservation in human myocardium. Biomed Biochim Acta. 1987;46(6):499-504. PMID 2890348
- [Background] Suleiman MS, Fernando HC, Dihmis WC, Hutter JA, Chapman RA. A loss of taurine and other amino acids from ventricles of patients undergoing bypass surgery. Br Heart J. 1993 Mar;69(3):241-5. doi: 10.1136/hrt.69.3.241. PMID 8461223
- [Background] Kimose HH, Ravkilde J, Helligso P, Knudsen MA, Thomassen AR, Nielsen TT, Djurhuus JC. Myocardial loss of glutamate after cold chemical cardioplegia and storage in isolated blood-perfused pig hearts. Thorac Cardiovasc Surg. 1993 Apr;41(2):93-100. doi: 10.1055/s-2007-1013829. PMID 8103947
- [Background] Smith RC, Leung JM, Mangano DT. Postoperative myocardial ischemia in patients undergoing coronary artery bypass graft surgery. S.P.I. Research Group. Anesthesiology. 1991 Mar;74(3):464-73. doi: 10.1097/00000542-199103000-00013. PMID 2001026
- [Background] Pisarenko OI, Lepilin MG, Ivanov VE. Cardiac metabolism and performance during L-glutamic acid infusion in postoperative cardiac failure. Clin Sci (Lond). 1986 Jan;70(1):7-12. doi: 10.1042/cs0700007. PMID 2867848
- [Background] Svedjeholm R, Ekroth R, Joachimsson PO, Ronquist G, Svensson S, Tyden H. Myocardial uptake of amino acids and other substrates in relation to myocardial oxygen consumption four hours after cardiac operations. J Thorac Cardiovasc Surg. 1991 Apr;101(4):688-94. PMID 2008107
- [Background] Svedjeholm R, Vanhanen I, Hakanson E, Joachimsson PO, Jorfeldt L, Nilsson L. Metabolic and hemodynamic effects of intravenous glutamate infusion early after coronary operations. J Thorac Cardiovasc Surg. 1996 Dec;112(6):1468-77. doi: 10.1016/S0022-5223(96)70005-3. PMID 8975838
- [Background] Vanhanen I, Hakanson E, Jorfeldt L, Svedjeholm R. Intravenous aspartate infusion after a coronary operation: effects on myocardial metabolism and hemodynamic state. Ann Thorac Surg. 1998 May;65(5):1296-302. doi: 10.1016/s0003-4975(98)00155-6. PMID 9594855
- [Background] Vanhanen I, Svedjeholm R, Hakanson E, Joachimsson PO, Jorfeldt L, Nilsson L, Vanky F. Assessment of myocardial glutamate requirements early after coronary artery bypass surgery. Scand Cardiovasc J. 1998;32(3):145-52. doi: 10.1080/14017439850140102. PMID 9764429
- [Background] Vanhanen I, Hakanson E, Jorfeldt L, Svedjeholm R. Myocardial uptake and release of substrates in patients operated for unstable angina: impact of glutamate infusion. Scand Cardiovasc J. 2003 May;37(2):113-20. doi: 10.1080/14017430310001230. PMID 12775312
- [Background] Svedjeholm R, Hakanson E, Szabo Z, Vanky F. Neurological injury after surgery for ischemic heart disease: risk factors, outcome and role of metabolic interventions. Eur J Cardiothorac Surg. 2001 May;19(5):611-8. doi: 10.1016/s1010-7940(01)00664-9. PMID 11343941
- [Background] Svedjeholm R, Hakanson E, Vanhanen I. Rationale for metabolic support with amino acids and glucose-insulin-potassium (GIK) in cardiac surgery. Ann Thorac Surg. 1995 Feb;59(2 Suppl):S15-22. doi: 10.1016/0003-4975(94)00917-v. PMID 7840694
- [Background] Rau EE, Shine KI, Gervais A, Douglas AM, Amos EC 3rd. Enhanced mechanical recovery of anoxic and ischemic myocardium by amino acid perfusion. Am J Physiol. 1979 Jun;236(6):H873-9. doi: 10.1152/ajpheart.1979.236.6.H873. No abstract available. PMID 443452
- [Background] Engelman RM, Rousou JA, Flack JE 3rd, Iyengar J, Kimura Y, Das DK. Reduction of infarct size by systemic amino acid supplementation during reperfusion. J Thorac Cardiovasc Surg. 1991 May;101(5):855-9. PMID 1673733
- [Background] Lazar HL, Buckberg GD, Manganaro AJ, Becker H, Maloney JV Jr. Reversal of ischemic damage with amino acid substrate enhancement during reperfusion. Surgery. 1980 Nov;88(5):702-9. PMID 7434210
- [Background] Bittl JA, Shine KI. Protection of ischemic rabbit myocardium by glutamic acid. Am J Physiol. 1983 Sep;245(3):H406-12. doi: 10.1152/ajpheart.1983.245.3.H406. PMID 6137148
- [Background] Haas GS, DeBoer LW, O'Keefe DD, Bodenhamer RM, Geffin GA, Drop LJ, Teplick RS, Daggett WM. Reduction of postischemic myocardial dysfunction by substrate repletion during reperfusion. Circulation. 1984 Sep;70(3 Pt 2):I65-74. PMID 6430593
- [Background] Pisarenko OI, Solomatina ES, Studneva IM, Ivanov VE, Kapelko VI, Smirnov VN. Protective effect of glutamic acid on cardiac function and metabolism during cardioplegia and reperfusion. Basic Res Cardiol. 1983 Sep-Oct;78(5):534-43. doi: 10.1007/BF01906464. PMID 6140002
- [Derived] Holm J, Vanky F, Svedjeholm R. Association of Glutamate Infusion With Risk of Acute Kidney Injury After Coronary Artery Bypass Surgery: A Pooled Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2024 Jan 2;7(1):e2351743. doi: 10.1001/jamanetworkopen.2023.51743. PMID 38252440
- [Derived] Jiang H, Holm J, Friberg O, Vanky F, Vidlund M, Tajik B, Yang Y, Svedjeholm R. Utility of NT-proBNP as an objective marker of postoperative heart failure after coronary artery bypass surgery: a prospective observational study. Perioper Med (Lond). 2021 Jul 13;10(1):21. doi: 10.1186/s13741-021-00194-4. PMID 34253255
- [Derived] Jiang H, Holm J, Vidlund M, Vanky F, Friberg O, Yang Y, Svedjeholm R. The impact of glutamate infusion on postoperative NT-proBNP in patients undergoing coronary artery bypass surgery: a randomized study. J Transl Med. 2020 May 11;18(1):193. doi: 10.1186/s12967-020-02351-7. PMID 32393387
- [Derived] Vidlund M, Tajik B, Hakanson E, Friberg O, Holm J, Vanky F, Svedjeholm R. Post hoc analysis of the glutamics-trial: intravenous glutamate infusion and use of inotropic drugs after cabg. BMC Anesthesiol. 2016 Aug 2;16(1):54. doi: 10.1186/s12871-016-0216-z. PMID 27484576
- [Derived] Holm J, Vidlund M, Vanky F, Friberg O, Hakanson E, Walther S, Svedjeholm R. EuroSCORE II and N-terminal pro-B-type natriuretic peptide for risk evaluation: an observational longitudinal study in patients undergoing coronary artery bypass graft surgery. Br J Anaesth. 2014 Jul;113(1):75-82. doi: 10.1093/bja/aeu088. Epub 2014 Apr 11. PMID 24727704
- [Derived] Holm J, Vidlund M, Vanky F, Friberg O, Hakanson E, Svedjeholm R. Preoperative NT-proBNP independently predicts outcome in patients with acute coronary syndrome undergoing CABG. Scand Cardiovasc J Suppl. 2013 Feb;47(1):28-35. doi: 10.3109/14017431.2012.731518. Epub 2012 Oct 10. PMID 22989031
- [Derived] Vidlund M, Holm J, Hakanson E, Friberg O, Sunnermalm L, Vanky F, Svedjeholm R. The S-100B substudy of the GLUTAMICS trial: glutamate infusion not associated with sustained elevation of plasma S-100B after coronary surgery. Clin Nutr. 2010 Jun;29(3):358-64. doi: 10.1016/j.clnu.2009.09.007. Epub 2009 Oct 22. PMID 19853332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 patients, 2 in each group were excluded because of intraoperative exclusion criteria
Period: Overall Study
Arm/Group | Intravenous Glutamate | Saline Infusion
Started | 430 | 435
Completed | 428 | 433
Not Completed | 2 | 2
Not completed — Intraoperative exclusion criteria | 1 | 1
Not completed — Intraoperative exclusion criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Glutamate | Saline Infusion | Total
Number analyzed (Participants) | 428 | 433 | 861
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 68 (9) | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 82 | 157
  Male | 353 | 351 | 704
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 428 | 433 | 861

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Perioperative Myocardial Infarction, Postoperative Heart Failure or Postoperative Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
Participants | 31 | 25

2. Secondary Outcome: Degree of Perioperative Myocardial Injury
Description: p-CK-MB postoperative day 1, p-troponin-T postoperative day 3
Time Frame: perioperative
Measure: Median (Inter-Quartile Range); unit: µg/L
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 411 | 427
µg/L
  CK-MB day 1 | 14 [10 to 23] | 14 [10 to 23]
  Troponin-T day 3 | 0.27 [0.16 to 0.57] | 0.24 [0.13 to 0.52]

3. Secondary Outcome: Postoperative Hemodynamic State
Description: Mixed venous oxygen saturation (SvO2) measured at weaning from cardiopulmonary bypass and on arrival to ICU
Time Frame: Until arrival to ICU
Measure: Mean (Standard Deviation); unit: percentage of saturated hemoglobin
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 416 | 421
percentage of saturated hemoglobin
  SvO2 at weaning from CPB | 72.0 (7.6) | 72.2 (7.3)
  SvO2 on arrival to ICU | 65.0 (7.0) | 64.9 (6.9)

4. Secondary Outcome: Postoperative Hemodynamic State in Patients With Severely Reduced Left Ventricular Ejection Fraction (LVEF<0.40)
Description: Hemodynamic instability despite inotropes or need for IABP at the end of surgery in patients with severely reduced left ventricular ejection fraction (LVEF<0.40)
Time Frame: End of surgery
Population: Moderately or severely reduced LVEF (<0.40)
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 71 | 75
Participants | 1 | 5

5. Secondary Outcome: Postoperative Renal Function
Description: maximum p-creatinine value recorded postoperatively < 30 days
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
µmol/L | 106 (50) | 106 (50)

6. Secondary Outcome: Number of Participants With Postoperative Stroke < 24 Hours
Description: Incidence of Postoperative stroke < 24 hours of surgery verifed by CT-scan
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
Participants | 4 | 6

7. Secondary Outcome: ICU Stay
Description: ICU duration of stay (hours)
Time Frame: ICU stay
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
hours | 21 [17 to 23] | 21 [17 to 23]

8. Secondary Outcome: Atrial Fibrillation
Description: Number of patients with atrial fibrillation recorded postoperatively
Time Frame: Hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
Participants | 147 | 152

9. Secondary Outcome: Severe Circulatory Failure in CCS Class IV Patients
Description: Severe circulatory failure according to prespecified criteria as judged by a blinded endpoints committee in CCS class IV patients
Time Frame: 30 days
Population: CCS class IV patients
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 225 | 233
Participants | 3 | 16

10. Secondary Outcome: 10-year Survival
Description: 10-year survival - related to intervention. Last follow-up August 3, 2022. Follow-up time ranged from 12.7-16.8 years.
Time Frame: 10 year - survival (crude)
Population: Two patients were lost to follow-up, one in each group. One patient had moved abroad, the other one for unknown reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 427 | 432
Participants | 301 | 301

11. Secondary Outcome: Postoperative Mortality
Description: Postoperative mortality within 30 days of surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate | Saline Infusion
Number analyzed (Participants) | 428 | 433
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality over a 10-year period. Serious and Other adverse events assessed over 30 days or in hospital
Description: All-cause mortality was monitored over a 10-year period. Serious and Other adverse events were monitored/assessed over 30 days or in hospital
Arm/Group | Intravenous Glutamate | Saline Infusion
All-Cause Mortality (participants affected / at risk) | 126/427 | 131/432
Serious Adverse Events (participants affected / at risk) | 54/428 | 59/433
Other Adverse Events (participants affected / at risk) | 164/428 | 165/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Glutamate (N=428) | Saline Infusion (N=433)
Stroke < 24 hours (Nervous system disorders) | 4 | 6 — Stroke within 24 hours of surgery
Severe circulatory failure (Cardiac disorders) | 10 | 18 — Postoperative heart failure according to prespecified criteria
Perioperative myocardial infarction (Cardiac disorders) | 11 | 6 — Troponin-T > 2.0 μg/L on the third or fourth postoperative day
Cardiac mortality (Cardiac disorders) | 1 | 4 — Death within 30 days or in hospital due to cardiac cause as determined by a blinded end-point committee
Postoperative dialysis (Renal and urinary disorders) | 2 | 6 — New onset dialysis postoperatively
Reoperation for bleeding (Blood and lymphatic system disorders) | 22 | 21 — Reoperation for bleeding during the postoperative course
Infection (Infections and infestations) | 4 | 8 — Infection requiring surgery (mainly deep sternal wound infections)
Postoperative mortality (Surgical and medical procedures) | 4 (4) | 5 (5) — All-cause mortality within 30 days of surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Glutamate (N=428) | Saline Infusion (N=433)
Postoperative nausea (Gastrointestinal disorders) | 139 | 114 — Postoperative nausea as reported by attending nurse
Postoperative atrial fibrillation (Cardiac disorders) | 147 | 152 — Postoperative atrial fibrillation recorded in the institutional database
Infection (Infections and infestations) | 33 | 27 — Postoperative infection not requiring surgery or extending hospital stay
Respiratory (Respiratory, thoracic and mediastinal disorders) | 39 | 45 — Respiratory problems (atelectasis, pleural effusion, respiratory discomfort, need for oxygen etc) reported but not extending hospital stay
Skin reaction (Skin and subcutaneous tissue disorders) | 3 | 7 — Rash, itching or other skin reaction reported by attending nurse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No